CLINICAL TRIAL: NCT00275223
Title: Insulin Resistance in Severely Obese Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: R03 DK67167 (completed); R03DK067167 (NIH)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Obesity; Insulin Resistance; Diabetes
Keywords: adipose tissue; adipocytokines
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study aims to understand the biological processes that link obesity to diseases including insulin resistance and diabetes. Our approach involves studying the health of patient undergoing weight loss either via weight reduction surgery or by medically supervised liquid formula diets. Patients must be enrolled in a weight treatment program at Emory Bariatrics, Emory University, Atlanta GA, to be eligible for this study. This study does not cover the cost of treatment at Emory Bariatrics. The hypothesis is that decreases in adipose-tissue derived factors during weight loss will be related to improvement in insulin function.

DETAILED DESCRIPTION:
Severe obesity affects 4.7% of the U.S. population. A significant number of these individuals suffer from impaired glucose tolerance and type II diabetes due to insulin resistance (IR). Although it is generally accepted that the accumulation of intraabdominal (IA) fat increases the risk of developing IR, the mechanisms responsible for this phenomenon are not yet understood. In addition, the role of subcutaneous (SC) fat towards the etiology of IR - protective, inert or detrimental - is still under debate. This is because SC adipose tissue releases adipocytokines (IL-6, leptin, TNF- ) that have been demonstrated to impair insulin action. In individuals who are severely obese, hyperinsulinemia may induce an exaggerated production of adipocytokines from IA compared to SC fat stores. Our specific aims are: (1) to determine relative contribution of abdominal SC fat versus IA fat to systemic levels of IL-6, leptin and TNF- in lean and in severely obese individuals; (2) to determine the effects of systemic adipocytokine concentrations on whole body as well as tissue sensitivity to insulin. Hypothesis: (a) In the context of severe obesity, IA fat produces increased quantities of IL-6, leptin and TNF- compared to SC fat; (b) In severely obese patients undergoing weight loss, whole body and tissue IR can be predicted by changes in systemic adipocytokines. Methods: Adipose tissue content of IL-6, leptin and TNF- will be determined by ELISA in biopsies obtained from IA and SC fat stores in lean and severely obese patients. Computer tomography-determined areas of IA and SC fat will be related to changes in systemic adipocytokines at baseline and 6-mo following weight loss therapy. Changes in systemic IL-6, leptin and TNF- will be assessed from measurements made at baseline and following 6-mo weight loss. For this time period we will also determine changes in whole body (via IVGTT) and tissue sensitivity to insulin (via glucose uptake into muscle and fat). Relationships between systemic adipocytokines and IR will be assessed using uni- and multivariate correlation analysis. These novel studies will determine whether hypersecretion of adipocytokines by IA versus SC adipose tissue induces IR in patients with severe obesity.

ELIGIBILITY:
Inclusion Criteria:

Enrolled in weight treatment program at Emory Bariatrics

Exclusion Criteria:

Male Smoker

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Nana Gletsu, Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Gletsu N, Lin E, Khaitan L, Lynch SA, Ramshaw B, Raziano R, Torres WE, Ziegler TR, Papanicolaou DA, Smith CD. Changes in C-reactive protein predict insulin sensitivity in severely obese individuals after weight loss surgery. J Gastrointest Surg. 2005 Nov;9(8):1119-26; discussion 1127-8. doi: 10.1016/j.gassur.2005.07.035. PMID 16269383